CLINICAL TRIAL: NCT04170218
Title: Quality of Care for Knee and Hip Osteoarthritis in Elderly Patients: a Multicentric Observational Study in France Using Quality Indicators Assessed by Questionnaire
Brief Title: Quality of Care for Knee and Hip Osteoarthritis in Elderly Patients
Acronym: QSAMISA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190201
Record Dates: First submitted 2019-10-25; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: Knee Osteoarthritis; Hip Osteoarthritis; Quality of Healthcare; Elderly
Keywords: knee osteoarthritis; hip osteoarthritis; quality of healthcare; elderly
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Hip and knee osteoarthritis (OA) was ranked in 2010 as the eleventh highest contributor to global disability. In France in 2014, non-spinal OA was the leading self-reported cause of morbidity among adults over sixty-five years of age, with a prevalence of 49.5 per cent. OA is known to be the first cause of disability in activities of daily life and a risk factor of frailty among people over seventy-five years of age. Despite its major impact on the elderly population's quality of life and health, quality of care for OA in elderly patients remains understudied.

Objective: The study aims to assess the quality of care for knee and hip OA in patients aged 75 years and over.

DETAILED DESCRIPTION:
Method: This prospective multicentric observational cohort study enrolls participants of 75 years and over with symptomatic hip or knee OA for more than three months, hospitalized in seven geriatric departments of three hospitals of "Assistance Publique - Hôpitaux de Paris", for any cause of admission. Quality of care for OA before hospitalization is assessed by the Assessing Care of Vulnerable Elderly's (ACOVE) quality indicators (QI) for OA, using a questionnaire. The primary endpoint is the pass rate for the ACOVE's QI about referral to an orthopedic surgeon for patients with severe functionally compromising knee or hip OA. The secondary endpoints are the pass rates for the six others ACOVE's QI for OA (annual assessment of functional status and degree of pain ; exercise therapy for patients with newly diagnosed knee OA ; education regarding the natural history, treatment, and self- management of OA ; acetaminophen as first-line pharmacologic therapy ; advising patients treated with non-steroidal anti-inflammatory drugs (NSAIDs) of their risks ; offering prophylaxis with a proton-pump inhibitor or misoprostol to patients treated with non-selective NSAIDs) and other elements of hip or knee OA care not assessed by the seven QI (including use of opioid analgesics, NSAIDs, intra-articular infiltrations, joint replacements). The sample is described with a rheumatologic assessment including Western Ontario and MACmaster universities osteoarthritis index (WOMAC) and Kellgren-Laurence classification, and with a geriatric assessment including nutritional status, Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) scores, Mini Mental State Examination (MMSE) score, Timed Up and Go walking test, modified Short Emergency Geriatric Assessment (mSEGA) scale and Cumulative Illness Rating Scale for Geriatrics (CIRS-G). Participants also complete the 12-Item Short Form Survey version 2 (SF-12v2) quality of life questionnaire. They receive a call twelve months after inclusion to collect vital status, orthopedic consultation and joint replacement during the last year.

ELIGIBILITY:
Inclusion Criteria:

* patients aged seventy-five years or over
* with symptomatic hip or knee osteoarthritis according to the American College of Rheumatology criteria
* with pain for more than three months
* affiliated to French social security
* having given their oral non-opposition to participate (or oral non-opposition of the guardian in case of legal guardianship)

Exclusion Criteria:

* clinical or radiological sign suggesting a differential diagnosis for hip or knee pain
* acute disease with clinical repercussion on walking
* life-threatened patients

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients hospitalized in seven geriatric departments of three hospitals of "Assistance Publique - Hôpitaux de Paris", for any cause of admission
Sampling Method: Probability Sample
Enrollment: 405 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
number of participants referred to an orthopedic surgeon as assessed by ACOVE's quality indicator questionnaire | at enrollment

SECONDARY OUTCOMES:
rate of eligible patients who passed the quality indicator about annual assessment of functional status and degree of pain, assessed by questionnaire | at enrollment
  The eligibility criterion is answer "yes" to the question "Do you have pain in your joints that bothers you a lot on most days?". The pass criterion is a "yes" response to either of the two questions "In the past 12 months, has any doctor or nurse asked you about the severity of your joint pain?" "In the past 12 months, has any doctor or nurse asked you if your joint pain affects the things you like or need to do?". The rate is calculated using the numerator as the number of eligible patients who passed the quality indicator and the denominator as the number of patients eligible for the quality indicator.
rate of eligible patients who passed the quality indicator about exercise therapy for patients with newly diagnosed knee osteoarthritis, assessed by questionnaire | at enrollment
  The eligibility criteria are knee pain that had lasted at least 3 months, health did not limit the patient's ability to bathe or dress, and patients or surrogates indicated that the patient did not have severe dementia. The pass criterion is a "yes" response to the question "Have you ever been sent to physical therapy or an exercise group or class for your knee pain?". The rate is calculated using the numerator as the number of eligible patients who passed the quality indicator and the denominator as the number of patients eligible for the quality indicator
rate of eligible patients who passed the quality indicator about education regarding the natural history, treatment, and self- management of osteoarthritis, assessed by questionnaire | at enrollment
  The eligibility criterion is pain in any joint lasting at least 6 months. The pass criterion is a a "yes" response to at least 1 of the 3 questions "Has any doctor or nurse ever talked to you about what your arthritis or joint pain will be like as time goes on, or the natural history of arthritis?" "Has any doctor or nurse ever talked to you about how to keep your arthritis or joint pain from getting worse?" "Has any doctor or nurse ever talked to you about how your arthritis can be treated?". The rate is calculated using the numerator as the number of eligible patients who passed the quality indicator and the denominator as the number of patients eligible for the quality indicator.
rate of eligible patients who passed the quality indicator about acetaminophen as first-line pharmacologic therapy, assessed by questionnaire | at enrollment
  The eligibility criterion is a "yes" response to the question "Has any doctor or nurse recommended any treatments for your joint pain?". The pass criterion is a "yes" response to the question "Did any doctor or nurse recommend you try acetaminophen before other medications for your joint pain?". Trade names of acetaminophen are mentioned to help participants. The rate is calculated using the numerator as the number of eligible patients who passed the quality indicator and the denominator as the number of patients eligible for the quality indicator.
rate of eligible patients who passed the quality indicator about advising patients treated with non-steroidal anti-inflammatory drugs (NSAIDs) of their risks, assessed by questionnaire | at enrollment
  The eligibility criteria are NSAID on medication list, or a "yes" response to the question "Do you take any medications like aceclofenac, celecoxib, diclofenac, etoricoxib, ibuprofene, indometacine, ketoprofene, naproxene or piroxicam ? These medications are known as non-steroidal anti-inflammatory drugs". Corresponding trade names are mentioned to help participants. The pass criterion is a "yes" response to the question "Did any doctor or nurse or pharmacist tell you about the possible side effects or risks from taking this medication?". The rate is calculated using the numerator as the number of eligible patients who passed the quality indicator and the denominator as the number of patients eligible for the quality indicator.
rate of eligible patients who passed the quality indicator about offering prophylaxis with a proton-pump inhibitor or misoprostol to patients treated with non-selective NSAIDs, assessed by questionnaire | at enrollment
  The eligibility criteria are NSAID on medication list, or a "yes" response to the question "Do you take any medications like aceclofenac, diclofenac, ibuprofene, indometacine, ketoprofene, naproxene or piroxicam?". Corresponding trade names are mentioned to help participants. The pass criterion is a "yes" response to the question "Did any doctor or nurse recommend you take another medication to protect your stomach or intestines or from developing an ulcer? For example omeprazole, esomeprazole, pantoprazole, lansoprazole or misoprostol". Corresponding trade names are mentioned to help participants. The rate is calculated using the numerator as the number of eligible patients who passed the quality indicator and the denominator as the number of patients eligible for the quality indicator.
percentage of patients taking non-steroidal anti-inflammatory drugs for their hip or knee osteoarthritis, assessed by questionnaire and reading current medical prescription | at enrollment
percentage of patients taking opioid analgesics for their hip or knee osteoarthritis, assessed by reading current medical prescription | at enrollment
percentage of patients taking symptomatic slow-acting anti-arthritics, assessed by assessed by reading current medical prescription | at enrollment
percentage of patients taking non-steroidal anti-inflammatory topically applied, assessed by assessed by reading current medical prescription | at enrollment
percentage of patients treated with intra-articular infiltration of corticosteroid, assessed by questionnaire | at enrollment
percentage of patients treated with intra-articular infiltration of visco-supplementation, assessed by questionnaire | at enrollment
percentage of patients who consulted a rheumatologist for their knee or hip osteoarthritis, assessed by questionnaire | at enrollment
percentage of patients who beneficiate from a modification of their medical prescription related to their knee or hip osteoarthritis treatment during or after their stay in the inclusion geriatric department, assessed by reading the medical record | after the patient discharge
percentage of patients referred to an orthopedic surgeon during or after their stay in the inclusion geriatric department, assessed by reading the medical record | after the patient discharge
percentage of patients referred to an orthopedic surgeon who really consulted the orthopedic surgeon, assessed by calling the patient one year after inclusion | one year after inclusion
percentage of patients referred to an orthopedic surgeon who beneficiated from a joint replacement for their hip or knee, assessed by calling the patient one year after inclusion | one year after inclusion
vital status at one year | one year after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe David, PhD, Study Director
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU HENRI MONDOR, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION